CLINICAL TRIAL: NCT03798145
Title: Surgical Retinotomy for the Treatment of Glaucoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49075
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Retinotomy (Experimental): Surgical retinotomy will be constructed in the area of the scotoma.
  Interventions: Procedure: Surgical Retinotomy

INTERVENTIONS:
Procedure: Surgical Retinotomy — Surgical removal of small areas of retinal to increase outflow through the posterior drainage pathway.

SUMMARY:
Glaucoma is a leading cause of blindness worldwide. It is caused by persistently elevated intraocular pressure causing progressive visual field loss. While a number of conventional medical and surgical therapies exist, a significant number of patients fail to respond resulting in persistently elevated intraocular pressure and eventual blindness. While outflow from the eye primarily occurs through the front of the eye, there is an often overlooked pathway to remove fluid that is beneath the retina. Surgical removal of retina to create paths for outflow (surgical retinotomy) in areas damaged by glaucoma can provide access to this alternative outflow pathway thereby reducing intraocular pressure and halting the vision loss.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate that focal surgical retinotomies (holes in the retina) can result in predictable and lasting reduction in intraocular pressure while eliminating the risks associated with surgical retinectomy (broad areas of retinal removal).

In the late 1990s and early 2000s, Joussen et al pioneered a technique to lower intraocular pressure in patients with advanced untreatable glaucoma. All patients had intraocular pressures on average above 40 that were unresponsive to any available treatments. Forty-four patients underwent broad areas of retinal removal (retinectomy). All patients exhibited dramatic reductions in intraocular pressure which were maintained for 5 years (Joussen 2003). Unfortunately, the technique carried significant risks. 1) a subset of patients had excessively low intraocular pressure reductions. 2) a subset of patients had secondary proliferative vitreoretinopathy (a scarring response) that resulting in retinal deatchment. Despite its incredible effectiveness, these risks made clinicians hesitant to adopt the technique. Additionally, glaucoma specialists are unable to perform the technical procedures required creating a chasm between diagnosing physician (glaucoma specialist) and the treating physician (retina specialist). Finally, surgical microtools tools at the time were still in their infancy.

The current proposal attempts to make critical modifications to the technique used by Joussen et al. (2003). First and foremost, we plan to use surgical retinotomies (holes in the retina) in lieu of a broad surgical retinectomy (broad peripheral retinal removal). This is a critical difference. Removal of the peripheral retina to the ora serrata carries significant risk of postoperative proliferative vitreoretinopathy. This is largely due to residual vitreous which cannot be removed from the far peripheral retina. This residual vitreous contracts in the postoperative period causing elevation of the retinectomy edges allowing for retinal detachment. Surgical retinotomies (holes in the retina), that do not involve the vitreous base are commonly used in retina surgery and do not carry anywhere close to the risk of retinal detachment that surgical retinectomy carries. As an example, the majority of retinal detachments are repaired by draining fluid through an iatrogenic surgical retinotomy (a hole created by the surgeon in the retina). These holes are created in the posterior retina and yet are virtually always undetectable by the patient. (Of note, a peripheral retinotomy is even harder to detect). More recently, there has been an upsurge of free-flap autologous retinal transplantation for macular holes (Grewal 2016) and macular degeneration (Parolini 2018). In these surgical procedures, an area of peripheral retina is removed and transplanted to the macula. The site of removal leaves a hole in the retina. In these studies the rate of redetachment in patients in whom a retinotomy was created is no higher than that of other standard retina surgeries. It is therefore clear that creation of retinal holes (retinotomy) is far different in terms of long-term risks than broad retinal removal to the ora serrata (retinectomy). Additionally, this increase in retina transplantation has been made possible by the microsurgical surgical tools that are now available. However, in the case of both the retinal detachment repair and autologous transplantation, the retinotomy size is not sufficient to induce intraocular pressure lowering effects. We therefore seek to build upon the original work from Joussen et al (2003) which showed that retina removal can have dramatic intraocular pressure lowering effects, but seek to use surgical retinotomies (holes in the retina) to achieve this retinal removal thereby avoiding his surgical complications while capitalizing on the long-term efficacy. By varying the size and number of surgical retinotomy, we will be able to provide a normogram for effective prediction of intraocular pressure lowering effects. By effectively predicting the magnitude of this surgical procedure, ophthalmologists will have a predictable and reliable method for treating glaucoma. Furthermore, because a surgical retinotomy does not close, it is predicted to provide a life-long effect.

ELIGIBILITY:
Inclusion Criteria:

Glaucoma with reproducible and progressive peripheral field loss Elevated Intraocular pressure despite topical medications and filtering surgery (trabeculectomy, tube shunts) Pseudophakia (prior cataract surgery) Greater than 50 years old

Exclusion Criteria:

Uveitic Glaucoma Foveal threatening visual field loss (field loss within 5 degrees of fixation) (i.e. advanced glaucoma) Active ophthalmic infection Monocular (functional vision in only one eye) Rapidly progressive glaucoma (as assessed by more than -1.00 MD drop over three months of visual field testing) Non-native English Speakers

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 2 years
  Percentage Reduction in Intraocular Pressure

SECONDARY OUTCOMES:
Visual Field Progression | 2 years
  Visual Field Progression on HVF 24-2 or Goldmann Visual Field

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grewal DS, Mahmoud TH. Autologous Neurosensory Retinal Free Flap for Closure of Refractory Myopic Macular Holes. JAMA Ophthalmol. 2016 Feb;134(2):229-30. doi: 10.1001/jamaophthalmol.2015.5237. No abstract available. PMID 26720054
- [Background] Joussen AM, Walter P, Jonescu-Cuypers CP, Koizumi K, Poulaki V, Bartz-Schmidt KU, Krieglstein GK, Kirchhof B. Retinectomy for treatment of intractable glaucoma: long term results. Br J Ophthalmol. 2003 Sep;87(9):1094-102. doi: 10.1136/bjo.87.9.1094. PMID 12928275
- [Background] Parolini B, Grewal DS, Pinackatt SJ, Baldi A, Di Salvatore A, Besozzi G, Finzi A, Cardillo D, Mahmoud TH. COMBINED AUTOLOGOUS TRANSPLANTATION OF NEUROSENSORY RETINA, RETINAL PIGMENT EPITHELIUM, AND CHOROID FREE GRAFTS. Retina. 2018 Sep;38 Suppl 1(Suppl 1):S12-S22. doi: 10.1097/IAE.0000000000001914. PMID 29210941
- [Background] Ramli N, Htoon HM, Ho CL, Aung T, Perera S. Risk factors for hypotony after transscleral diode cyclophotocoagulation. J Glaucoma. 2012 Mar;21(3):169-73. doi: 10.1097/IJG.0b013e318207091a. PMID 21336153
- [Background] Jain K, Dubey S, Pegu J. Comparison of Efficacy and Complications of Cyclophotocoagulation and Second Glaucoma Drainage Device After Initial Glaucoma Drainage Device Failure. J Glaucoma. 2018 Aug;27(8):e140. doi: 10.1097/IJG.0000000000000955. No abstract available. PMID 29578892